CLINICAL TRIAL: NCT03678428
Title: FUDR/Oxaliplatin HAI Plus Irinotecan Chemotherapy vs. FOLFOXIRI Chemotherapy in Treating Initially Unresectable CRCLM
Brief Title: FUDR/Oxaliplatin HAI Plus Irinotecan vs. FOLFOXIRI Chemotherapy in Treating Initially Unresectable CRCLM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Production halt of FUDR in China
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Director, Department of Medical Oncology, Principal Investigator, Clinical Professor, Yuhong Li, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIUMPH
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Floxuridine; Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FUDR/Oxaliplatin HAI plus irinotecan (Experimental): Patients will receive Systemic CPT-11 + HAI (FUDR+L-OHP) every 28 days:
  Irinotecan 150 mg/m2 IV over 90 minutes on Day 1; followed by Oxaliplatin 85 mg/m2 over 3 hours through the HAI pump on Day 1 and 0.12 mg/kg/day floxuridine (FUDR) and 25 mg dexamethasone in normal saline to a total volume of 300 ml will be administered through the HAI pump.
  then Irinotecan 150 mg/m2 IV over 90 minutes on Day 15, followed by Oxaliplatin 85 mg/m2 IV over 3 hours on Day 15.
  This will be repeated on Day 1 of each 28-day cycle. FUDR will be administered through a 14-day continuous infusion with the HAI pump.
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin HAI; Drug: Floxuridine
- FOLFOXIRI (Active Comparator): Patients will receive Systemic FOLFOXIRI every 28 days:
  Irinotecan 150 mg/m2 IV over 90 minutes on Day 1 and Day 15; Oxaliplatin 85 mg/m2 IV in 3-6 hours on Day 1 and Day 15; Leucovorin 200mg/m2 and 5-FU 2400mg/m2 CIV in 46 hours on Day 1 and Day 15.
  Interventions: Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 150 mg/m2 IV over 90 minutes on Day 1 and 15.
Drug: Oxaliplatin HAI — Oxaliplatin 85 mg/m2 over 3 hours will be administered through the HAI pump on day 1. Oxaliplatin 85 mg/m2 IV over 3 hours on day 15.
  Arms: FUDR/Oxaliplatin HAI plus irinotecan
Drug: Floxuridine — 0.12 mg/kg/day floxuridine (FUDR) and 25 mg dexamethasone in normal saline to a total volume of 300 ml will be administered through the HAI pump.
  Arms: FUDR/Oxaliplatin HAI plus irinotecan
Drug: Leucovorin — Leucovorin 200mg/m2 IV on Day 1 and 15.
  Arms: FOLFOXIRI
Drug: 5-FU — 5-FU 2400mg/m2 CIV in 46h on Day 1 and 15.
  Arms: FOLFOXIRI
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 IV over 3 hours on Day1 and 15.
  Arms: FOLFOXIRI

SUMMARY:
The aim of the trial is to compare the objective response rates of FUDR/Oxaliplatin HAI plus CPT-11 and FOLFOXIRI chemotherapy in patients with initially non-resectable metastatic colorectal cancer liver metastases. The patients will be treated with systemic FOLFOXIRI chemotherapy or FUDR/Oxaliplatin hepatic arterial infusion with CPT-11 systemic chemotherapy.

DETAILED DESCRIPTION:
Previous studies and our experience have proved the efficacy and safety of systemic chemotherapy combined with hepatic arterial infusion (HAI) with floxuridine and dexamethasone in patients with initially unresectable colorectal liver metastasis. Hepatic arterial infusion oxaliplatin trials have been done with oxaliplatin alone and in combination with irinotecan, 5-FU/LV, and mitomycin-C and have showed that Hepatic arterial infusion oxaliplatin and FUDR could increase response rate and resection rate for colorectal liver metastasis. Therefore, we designed this study to compare objective response rates of FUDR/Oxaliplatin HAI plus CPT-11 and FOLFOXIRI chemotherapy in patients with initially non-resectable metastatic colorectal cancer liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤70.
* Diagnosed as colorectal adenocarcinoma by histology.
* Confirmed as liver metastases by medical imaging or pathology.
* MDT determined as unresectable liver metastases, defined as:①more than 5 metastases; ②unable to conduct R0 resection; ③no sufficient residual liver volume after resection; ④none of 3 hepatic vein can be reserved after resection, no sufficient blood supply or bibliary duct can be reserved, none of 2 adjacent liver segment can be reserved. Whenever meets any of the criteria mentioned above would be defined as unresectable liver metastases.
* No previous treatment aiming at treating liver metastases, including chemotherapy, surgery, radiotherapy, transcatheter hepatic arterial chemoembolization(TACE) or target therapy.
* Confirmed by CT, MRI or PET/CT(if necessary) that there is no extrahepatic metastases or only oligos extrahepatic metastases(no more than 2 organs and 5 leisions, maximum diameters of single leision ≤ 1cm).
* Unsuitable for cetuximab treatment(RAS mutation, unable to afford the cost).
* No hematologic dysfunction(Platelets >90×10^9/L; WBC >3×10^9/L; Neutrophil >1.5×109/L).
* Serum bilirubin ≤ 1.5 × ULN; aminotransferase ≤ 5 × ULN.
* No ascites; no coagulation dysfunction; albumin ≥ 30g/L.
* Hepatic function was classified as class A by Child-Pugh classification.
* Serum creatinine < 1 × ULN, or creatinine clearance rate(CCR) > 50ml/min(calculated by Cockcroft-Gault formula).
* ECOG scored as 0-1.
* Life expectancy > 3 months.
* Informed consent.
* Willing and able to receive follow-up until death or trial is finished or trial is terminated.

Exclusion Criteria:

* Presence of extensive extrahepatic metastases(more than 2 organs and 5 leisions, or maximum diameter of single leision > 10 cm).
* Severe arterial embolism or ascites.
* Presence of hemorrhagic tendency or coagulation dysfunction.
* Presentive of hypertensive crisis or hypertensive encephalopathy.
* Severe uncontrolled systemic complications, such as infection or diabetes.
* Severe clinical CVD(cardiovascular disease), such as cerebrovascular accident(within 6 months before recruitment), myocardial infarction(within 6 months before recruitment), uncontrolled hypertension; unstable angina pectoris; congestive heart-failure(NYHA 2-4 grade); arrhythmia that needs medication treatment.
* Previous diagnosed or physical examination showed presence of central nervous system(CNS) disease(i.e. primary brain tumor, epilepsy uncontrolled by standard treatment, any history of brain metastases or stroke).
* Previous history of other malignancy within 5 years(except basal cell carcinoma after radical resection and/or cervical carcinoma in situ).
* Received any medication under research within 28 days before the trial.
* Any residual toxicity of previous chemotherapy(except hair loss), i.e. peripheral neuropathy ≥ NCI CTC v3.0 Grade 2, will be excluded from oxaliplatin-based chemotherapy regimen research pair.
* Allergic to any medication involved in the trial.
* Pregnant and lactating women.
* Patient who does not use or refuses to take any appropriate contraceptive measures (intrauterine contraceptive ring, barrier contraception combined with spermicidal gel or sterilization operation), including women of childbearing age (within 2 years after the last menstrual period) and men who are with possible fertility.
* Unable or unwilling to comply with the research plan.
* The existence of any other disease, dysfunction caused by metastatic lesions, or suspicious disease found on the regular examination, which indicating contraindications to the use of study drugs or may bring high risks of treatment related complications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate and bilateral 95% confidence interval | Up to 2-4 months
  defined as complete remission rates and partial remission rates after treatment.

SECONDARY OUTCOMES:
R0 resection rates | Up to 2-4 months
  defined as no macroscopic or microscopic residual tumor
Depth of tumor regression(DpR) | Up to 2-4 months
  defined as the largest depth of tumor regression
Progress-free Survival(PFS) | Up to 2-4 months
  defined as the period from the date of receiving treatment to disease progress caused by any reason.
Relapse-free Survival(RFS) of patients with resectable tumor | Up to 2-4 months
  defined as the period from the date of resection to tumor relapse caused by any reason.
Overall Survival(OS) | Up to 2-4 months
  defined as the period from the date of receiving treatment to death caused by any reason.
Adverse events, servere adverse events and surgery-related adverse events rates | Up to 2-4 months
  defined as the incidence and severity of adverse events related to chemotherapy, HAI and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhong Li, MD, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China